CLINICAL TRIAL: NCT01346826
Title: Safety of Accelerated Infliximab Infusions in Patients With Inflammatory Bowel Disease: A Prospective, Randomized, Double-Blind, Controlled Trial
Brief Title: Safety of Accelerated Infliximab Infusions in Patients With Inflammatory Bowel Disease (IBD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Suk-Kyun Yang, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-0181
Record Dates: First submitted 2011-05-02; First posted 2011-05-03 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: Crohn's disease; Ulcerative colitis; Infliximab; Infusion reaction
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2 hours-infusion group (Active Comparator): Number of patients: 57 (Standard 2 hours-infusion group)
  Interventions: Drug: Standard 2 hours-infusion
- 1 hour-infusion group (Experimental): Number of patients: 59 (1 hour-infusion group)
  Interventions: Drug: Accelerated 1 hour-infusion
- 30 minutes-infusion group (Experimental): Number of patients: 59 (30 minutes-infusion group)
  Interventions: Drug: Accelerated 30 minutes-infusion

INTERVENTIONS:
Drug: Standard 2 hours-infusion — Patients without any infusion reactions during more than 4 infusions for 2 hours are randomized to one of three study groups.
  After randomization to 2 hours-infusion group, patients get 5 mg/kg infliximab infusion for 2 hours. Total infusion number after randomization is 7.
  Other Names: Infliximab (Remicade, Centocor, Malvern, Philadelphia, PA)
  Arms: 2 hours-infusion group
Drug: Accelerated 1 hour-infusion — Patients without any infusion reactions during more than 4 infusions for 2 hours are randomized to one of three study groups.
  After randomization to 1 hour-infusion group, patients get 5 mg/kg infliximab infusion for 1 hour. Total infusion number after randomization is 7.
  Other Names: Infliximab (Remicade, Centocor, Malvern, Philadelphia, PA)
  Arms: 1 hour-infusion group
Drug: Accelerated 30 minutes-infusion — Patients without any infusion reactions during more than 4 infusions for 2 hours are randomized to one of three study groups.
  After randomization to 30 minutes-infusion group, patients get 5 mg/kg infliximab infusion for 1 hour. If any infusion reactions do not develop during 2 infusions for 1 hour, patients get further 5 mg/kg infliximab infusion for 30 minutes. The total number of 30 minutes-infusion is 5.
  Other Names: Infliximab (Remicade, Centocor, Malvern, Philadelphia, PA)
  Arms: 30 minutes-infusion group

SUMMARY:
This study aims to test the hypothesis that the accelerated infusion of infliximab is not inferior to the conventional 2 hour infusion with respect to the frequency of infusion reaction.

DETAILED DESCRIPTION:
The standard protocol of infliximab administration is the infusion for 2 hours. However, due to the discomfort of patients and limitation of medical resources, the accelerated infusion is more desirable if accelerated infusion does not increase the frequency of infusion reaction. Recent observational studies showed that the accelerated infusion of infliximab for 1 hour or 30 minutes did not increase the frequency of infusion reaction if patients had not shown infusion reactions during previous 4 infusions for 2 hours. However, there are no randomized trials comparing the safety of accelerated infusion protocol and standard infusion protocol yet.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving infliximab for Crohn's disease or ulcerative colitis
* Ethnicity: Korean
* Patients who did not show any infusion reactions during 4 times of infliximab (5mg/kg) infusions for 2 hours
* Informed consents

Exclusion Criteria:

* Sever cardiopulmonary diseases
* Allergic diseases

  * Bronchial asthma
  * Allergic rhinitis
  * Atopic dermatitis
  * Other allergic diseases determined not suitable for study participation by investigators
* Severe liver disease
* Severe renal disease
* Body weight over 100 kg
* Other medical or surgical disease determined not suitable for study participation by investigators

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2011-05; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Total numbers of infusion reactions related with infliximab infusion | Within14 days after infliximab infusion
  Total numbers of infusion reactions (including acute and delayed reactions) related with infliximab infusion

SECONDARY OUTCOMES:
Numbers of severe infusion reactions related with infliximab infusion | Within14 days after infliximab infusion
  Numbers of severe infusion reactions (Systolic blood pressure < 80 mmHg with severe symptoms and signs necessiating stopping of infliximab infusion) related with infliximab infusion

CONTACTS AND LOCATIONS:
Overall Officials: Suk-Kyun Yang, MD, PhD, Principal Investigator — Department of Gastroenterology, Asan Medical Center, University of Ulsan College of Medicine
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clare DF, Alexander FC, Mike S, Dan G, Allan F, Lisa W, Peter HJ. Accelerated infliximab infusions are safe and well tolerated in patients with inflammatory bowel disease. Eur J Gastroenterol Hepatol. 2009 Jan;21(1):71-5. doi: 10.1097/MEG.0b013e3283081afe. PMID 19060632
- [Background] Van Assche G, Vermeire S, Noman M, Amant C, Weyts E, Vleminckx A, Vermeyen MJ, Rutgeerts P. Infliximab administered with shortened infusion times in a specialized IBD infusion unit: a prospective cohort study. J Crohns Colitis. 2010 Sep;4(3):329-33. doi: 10.1016/j.crohns.2009.12.012. Epub 2010 Jan 18. PMID 21122522
- [Background] Bhat S, Sharma D, Doherty P, Tham TC, Caddy GR. Are accelerated infliximab infusions safe in patients with inflammatory bowel disease? Inflamm Bowel Dis. 2010 Nov;16(11):1922-5. doi: 10.1002/ibd.21279. PMID 20848465
- [Background] Breynaert C, Ferrante M, Fidder H, Van Steen K, Noman M, Ballet V, Vermeire S, Rutgeerts P, Van Assche G. Tolerability of shortened infliximab infusion times in patients with inflammatory bowel diseases: a single-center cohort study. Am J Gastroenterol. 2011 Apr;106(4):778-85. doi: 10.1038/ajg.2011.61. Epub 2011 Mar 15. PMID 21407184